CLINICAL TRIAL: NCT06818500
Title: Resting Indicators of Vascular Health and Cardiovascular Reactivity in Females with "Normal-Weight Obesity"
Brief Title: Effects of Body Composition on Vascular Health in Females with a Healthy Body Weight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ball State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2201237-1
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Normal-weight Obesity; BMI; Stress
Keywords: BMI; Stress; Healthy BMI

STUDY DESIGN:
Intervention Model Description: We are studying human physiology of cardiovascular health in females with a normal BMI. We will not be using any drug interventions. Instead, participants will eat a high-fat meal at one visit and complete a stress task at the other visit. Vascular responses will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-fat meal trial (Experimental): During the "High-fat meal trial", participants will report fasted and consume two Jimmy Dean's breakfast bowls.
  Interventions: Other: high-fat meal
- Stress trial (Experimental): During the "Stress trial", participants will report fasted and undergo a stress task where they may experience mental stress.
  Interventions: Other: Stress

INTERVENTIONS:
Other: high-fat meal — Participants will report fasted and consume two Jimmy Dean breakfast bowls (sausage).
  Arms: High-fat meal trial
Other: Stress — Participants will report fasted and undergo a mental stress task.
  Arms: Stress trial

SUMMARY:
Most of the time, body weight is evaluated by looking at the ratio of your weight to your height. This measurement is called body mass index or BMI. However, BMI does not account for what your body is actually made up of (e.g., body fat versus muscle), which may be more important for determining cardiovascular disease risk. The investigators aim to understand vascular health in females with a "healthy" BMI with differing amounts of body fat and muscle mass. We will have participants come to the lab for two different study visits. At one visit, participants will eat a meal high in fat, and at the other visit, participants will undergo a stress task.

DETAILED DESCRIPTION:
The investigators will recruit females with a BMI in the normal (18.5-24.9 kg/m2) from the Ball State University campus and surrounding communities. Each participant will complete a meal trial and a stress trial in a randomized crossover design. At the meal trial, an intravenous catheter will be inserted and baseline blood sample collected. Then vascular measurements (i.e., flow-mediated dilation, pulse wave analysis, pulse wave velocity) will be performed. Each time vascular measurements are performed, the participants will lie in a quiet area to acclimate prior to beginning. Next, participants will consume a high-fat, Western style meal consisting of two Jimmy Deans Breakfast Bowls (sausage; 68 g fat; 880 kcal). Following completion of the meal, blood samples will also be collected 1, 2, 3, and 4 hours after the meal. Vascular measurements will be repeated 2 and 4 hours after the meal. Blood will be collected and stored as serum in order to measure triglycerides, HDL-C, and intestinal permeability (e.g., lipopolysaccharide binding protein) using commercially available ELISAs.

At the stress trial, an intravenous catheter will be inserted and baseline blood sample collected. Then vascular measurements (i.e., flow-mediated dilation, pulse wave analysis, pulse wave velocity) will be performed. Each time vascular measurements are performed, the participants will lie in a quiet area to acclimate prior to beginning. Next, participants will undergo the stress task. Then, blood samples will be collected at 10, 60, and 90 minutes after the stress task. Blood will be collected and stored as serum in order to measure epinephrine and inflammatory markers. Vascular measurements will also be repeated 10 and 90 minutes after the stress task.

ELIGIBILITY:
Inclusion Criteria:

* You are 18-50 years old
* Your biological sex is female
* BMI is in "normal" category (18.5-24.9 kg/m2) - this BMI requirement is due to our research aims
* You are not pregnant or expecting to become pregnant
* You are not postmenopausal
* You have not been diagnosed with a cardiometabolic condition (e.g., cardiovascular disease, type 2 diabetes)
* You have not been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* You do not regularly take anti-inflammatory drugs (more than 2x week) or are able to temporarily suspend use of anti-inflammatory drugs.
* You do not use lipid-lowering drugs (e.g., statins), glucose-lowering drugs (e.g., metformin) tobacco products, or any illicit drugs
* You do not have a pacemaker.
* You do not have dietary restrictions prohibiting you from eating the provided meal (e.g., vegan/vegetarian diets, gluten-free diet, relevant food allergies).
* You are able to stay in the supine position in the dark for at least 10 minutes

Exclusion Criteria:

* You are not 18-50 years old
* Your biological sex is not female
* Your BMI is not in the "normal" category (18.5-24.9 kg/m2) - this BMI requirement is due to our research aims
* You are pregnant or expecting to become pregnant (females only)
* You are postmenopausal
* You have been diagnosed with a cardiometabolic condition (e.g., cardiovascular disease, type 2 diabetes)
* You have been diagnosed with a chronic inflammatory condition (e.g., rheumatoid arthritis, inflammatory bowel disease).
* You regularly take anti-inflammatory drugs (more than 2x week) or are unable to temporarily suspend use of anti-inflammatory drugs.
* You use lipid-lowering drugs (e.g., statins), glucose-lowering drugs (e.g., metformin) tobacco products, or any illicit drugs
* You have a pacemaker.
* You do have dietary restrictions prohibiting you from eating the provided meal (e.g., vegan/vegetarian diets, gluten-free diet, relevant food allergies).
* You are unable to stay in the supine position in the dark for at least 10 minutes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Flow-mediated dilation | Through study completion, up to 1 year.
  The investigators will measure FMD at baseline, 2-hours, and 4-hours after meal trial. The investigators will measure FMD at baseline, post-stress task, and 90-minutes after the stress task.
Pulse wave analysis | Through study completion, up to 1 year.
  The investigators will measure PWA (i.e., augmentation index, augmentation index normalized to a heart rate of 75bpm, aortic/peripheral blood pressure) at baseline, 2-hours, and 4-hours after meal trial using Sphygmacor Xcel System. The investigators will measure PWA at baseline, post-stress task, and 90-minutes after the stress task.
Pulse wave velocity | Through study completion, up to 1 year.
  The investigators will measure PWV at baseline, 2-hours, and 4-hours after meal trial using the Sphygmacor Xcel System. The investigators will measure PWV at baseline, post-stress task, and 90-minutes after the stress task.

SECONDARY OUTCOMES:
Serum high-density lipoprotein cholesterol (HDL-C) | Through study completion, up to 1 year.
  The investigators will measure HDL-C at baseline and 1, 2, 3, and 4 hours after the meal. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum triglycerides | Through study completion, up to 1 year.
  The investigators will measure triglycerides at baseline and 1, 2, 3, and 4 hours after the meal. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum soluble CD14 (sCD14) | Through study completion, up to 1 year.
  The investigators will measure serum sCD14 at baseline and 1-, 2-, 3-, and 4-hours after the meal. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum lipopolysaccharide binding protein (LBP) | Through study completion, up to 1 year.
  The investigators will measure serum LBP at baseline and 1-, 2-, 3-, and 4-hours after the meal. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum epinephrine | Through study completion, up to 1 year.
  The investigators will measure serum epinephrine at baseline and 10-, 60- and 90-minutes after the stress task. Serum will be banked from each visit and this measurement will take place upon study completion.
Serum interleukin-6 (IL-6) | Through study completion, up to 1 year.
  The investigators will measure serum IL-6 at baseline and 1-, 2-, 3-, and 4-hours after the meal and 10, 60, and 90 minutes after the stress task. Serum will be banked from each visit and this measurement will take place upon study completion.
Heart rate variability (HRV) | Through study completion, up to 1 year.
  The investigator will analyze HRV pre-, during, and post-stress task during the stress trial (Task Force Monitor).
Beat-to-beat systolic and diastolic blood pressure (SBP/DBP) | Through study completion, up to 1 year.
  The investigator will analyze SBP/DBP pre, during, and post-stress task during the stress trial (Task Force Monitor).

OTHER OUTCOMES:
Body composition | Through study completion, up to 1 year.
  The investigators will measure body composition using dual energy x ray absorptiometry (DXA).
Systolic and diastolic blood pressure | Through study completion, up to 1 year.
  The investigators will measure blood pressure using an automated cuff (Omron).

CONTACTS AND LOCATIONS:
Locations (1):
- Ball State University- Nutrition Assessment Lab, Muncie, Indiana, United States

IPD SHARING:
Plan to Share IPD: No